CLINICAL TRIAL: NCT06848036
Title: Effectiveness of a Smart Community- and Home-based Integrated Care Services System for Elderly People in Rural Chinese Communities: A Randomized Controlled Trial in Changsha County
Brief Title: Effectiveness of a Smart Community- and Home-based Integrated Care Services System for Elderly People
Acronym: ESCHIC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Liu Zhihan (Other)
Responsible Party: Sponsor-Investigator, Liu Zhihan, Principal Investigator, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 234083; Self-funded (Other Grant/Funding Number: Liu Zhihan)
Record Dates: First submitted 2025-02-12; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Smart Community- and Home-based Integrated Care Services
Keywords: Integrated Care Services

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Receiving integrated care services through the "Hunan Province Medical Elderly Integration Intelligent Service Platform".
  Interventions: Behavioral: smart integrated care services
- Control group (No Intervention): Receive regular community care services, with no intervention, as a blank control

INTERVENTIONS:
Behavioral: smart integrated care services — Provide integrated care services through the 'Hunan Province Integrated Healthcare and Elderly Care Intelligent Service Platform,' including home-based care, mobile medical visits, and remote diagnosis and treatment services."
  Arms: Experimental group

SUMMARY:
In recent years, the widespread application of emerging information technologies such as artificial intelligence, the Internet of Things, big data, cloud computing, and 5G has made "smart " a new breakthrough in the integrated healthcare and elderly care model. Smart Community- and Home-based Integrated Care Services , utilizing methods such as home hospital beds and mobile medical visits, ensure that key elderly groups with disabilities, dementia, chronic diseases, advanced age, and disabilities can receive the necessary medical services at home. This not only allows the elderly to live in familiar home environments, maintaining their independence and dignity, but also alleviates the pressure on medical resources, enabling more resources to be allocated to emergency care and highly specialized nursing. However, the smart healthcare and elderly care platform model is still in the pilot stage and requires more scientific evidence to verify its actual impact on the health of the elderly.

The purpose： The purpose of this clinical trial is to understand and verify the potential health improvement effects of the smart healthcare and elderly care platform on the elderly. By collecting health indicator data at different time points before and after the intervention, the study will compare the differences in health indicators between community-dwelling elderly who have used the smart healthcare and elderly care platform and those who have not, providing scientific evidence for the promotion of the smart healthcare and elderly care platform model and further facilitating its application and popularization among the elderly in the community.

The main question it aims to answer is: Are community-dwelling elderly who use the smart healthcare and elderly care platform healthier than those who do not use the service? Participants will： Participants will be randomly divided into an experimental group and a control group. The elderly in the experimental group will use the "Hunan Province Integrated Healthcare and Elderly Care Intelligent Service Platform," while the control group will not use the platform for blank control.

Data collection： The research team will collect health indicator data four times, including SF-36, Activities of Daily Living (ADL), and the Geriatric Depression Scale (GDS), at baseline, 3 months post-intervention, 6 months post-intervention, and 12 months post-intervention.

DETAILED DESCRIPTION:
I. Recruitment Phase:

The study will recruit participants from Guoyuan Town, Changsha County. Eligible elderly individuals from rural communities will undergo qualification assessment based on inclusion/exclusion criteria. Accounting for a 20% attrition rate, the study plans to enroll 64 elderly participants from rural communities in Guoyuan Town.

II. Intervention Allocation Phase:

Participants will be randomly assigned to either the experimental or control group using computer-generated randomization. Baseline measurements will be collected using:

SF-36 Health Survey

Activities of Daily Living (ADL) scale

Geriatric Depression Scale (GDS)

The experimental group will receive integrated care services through the "Hunan Province Integrated Smart Healthcare and Elderly Care Service Platform", while the control group will receive standard community care. The intervention includes:

Educational seminars introducing "Hunan Province Integrated Smart Healthcare and Elderly Care Service Platform" services

Assistance with platform registration for experimental group participants

Implementation of integrated care services via the platform

III. Follow-up Phase:

Three follow-up assessments will be conducted at:

3 months post-intervention

6 months post-intervention

12 months post-intervention

Follow-up assessments will repeat baseline measurements (SF-36, ADL, GDS) to evaluate health status changes. Participant attrition will be documented through follow-up tracking. All data will undergo double-entry verification using two independent data clerks maintaining separate files, with regular cross-verification and final reconciliation after the last follow-up.

IV. Analysis Phase:

Statistical comparisons between groups will be performed using:

Independent t-tests

Analysis of variance (ANOVA)

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged ≥60 years
2. Normal verbal communication abilities
3. No self-reported visual or auditory impairments
4. Presence of a long-term, fixed caregiver who accompanies and lives with the participant
5. Both the participant and their family members are informed and consent voluntarily to participate in this study

Exclusion Criteria

1. Participants aged <60 years
2. Individuals suffering from severe physical or mental illnesses
3. Elderly individuals who have participated in other similar studies within the past year
4. Elderly individuals residing in institutions

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-08-07 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
SF-36 scale (Short Form 36 Health Survey) | Measurements were taken to obtain data after interventions at three months, six months, and twelve months.
  The SF-36 (Short Form 36 Health Survey) is a tool used to assess health-related quality of life across 8 dimensions, each scored from 0 to 100. A higher score indicates better health. The 8 dimensions are:
  Physical Functioning (PF): Ability to perform physical activities. Role-Physical (RP): Limitations due to physical health. Bodily Pain (BP): Pain intensity and impact. General Health (GH): Overall health perception. Vitality (VT): Energy levels and fatigue. Social Functioning (SF): Impact on social activities. Role-Emotional (RE): Limitations due to emotional problems. Mental Health (MH): Psychological well-being. Scores are calculated based on responses, with 0 representing the worst health and 100 the best. The higher the total score, the better the health.

SECONDARY OUTCOMES:
ADL scale（（Activity of Daily Living） | Measurements were taken to obtain data after interventions at three months, six months, and twelve months.
  ADL (Activities of Daily Living) is used to assess an individual's ability to perform basic activities of daily living, particularly self-care functions.The score for each option in the scale will be reported, with the minimum score for each option being 0 and the maximum score being 3. The scores will then be summed, with the total score having a minimum value of 0 and a maximum value of 20.Total possible scores range from 0 - 20, with lower scores indicating increased disability. If used to measure improvement after rehabilitation, changes of more than two points in the total score reflect a probable genuine change, and change on one item from fully dependent to independent is also likely to be reliable.
GDS scale（Geriatric Depression Scale) | Measurements were taken to obtain data after interventions at three months, six months, and twelve months.
  The GDS will evaluate the mental status of the elderly, using a questionnaire format.The GDS scale contains 15 items, and participants answer with "Yes" or "No." Each "Yes" is scored 1 point, and each "No" is scored 0 points. The total score is the sum of the individual item scores. A higher total score indicates more pronounced depressive symptoms. A score of ≥6 points suggests the presence of depressive mood, 0-5 points indicates no depressive mood, 6-9 points indicates mild depressive mood, and 10-12 points indicates severe depressive mood.

CONTACTS AND LOCATIONS:
Overall Officials: Zhihan Liu, Principal Investigator — School of Public Administration, Central South University
Locations (1):
- Changsha County Guoyuan Town Health Center, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Z, Wei H, Liu Z. Older Adults' Demand for Community-Based Adult Services (CBAS) Integrated with Medical Care and Its Influencing Factors: A Pilot Qualitative Study in China. Int J Environ Res Public Health. 2022 Nov 11;19(22):14869. doi: 10.3390/ijerph192214869. PMID 36429594
- [Background] Liu Z, Ouyang C, Gu N, Zhang J, He X, Feng Q, Chang C. Service quality evaluation of integrated health and social care for older Chinese adults in residential settings based on factor analysis and machine learning. Digit Health. 2024 Dec 19;10:20552076241305705. doi: 10.1177/20552076241305705. eCollection 2024 Jan-Dec. PMID 39711744
- [Background] Wang Z, Liu Z. Latent classes and related predictors of demand for home-and community-based integrated care for older Chinese adults. Front Public Health. 2023 Jun 23;11:1109981. doi: 10.3389/fpubh.2023.1109981. eCollection 2023. PMID 37427265
- [Background] Zhang W, He X, Liu Z. Factors and Mechanism Influencing Client Experience of Residential Integrated Health and Social Care for Older People: A Qualitative Model in Chinese Institutional Settings. Int J Environ Res Public Health. 2023 Mar 6;20(5):4638. doi: 10.3390/ijerph20054638. PMID 36901645

DOCUMENTS (3):
  • Study Protocol (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT06848036/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT06848036/SAP_001.pdf
  • Informed Consent Form (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT06848036/ICF_002.pdf